CLINICAL TRIAL: NCT03157050
Title: Intravenous Iron May Increase Depression Among Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Collaborators: New Jeddah Clinic Hospital (Industry)
Responsible Party: Principal Investigator, Mahmoud Hamada imam, Lecturer of Internal Medicine - Faculty of Medicine, Benha University
Other Study IDs: BN-13058
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Depression; Hemodialysis Complication; Iron Deficiency Anemia
MeSH Terms: conditions — Depression; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intravenous iron therapy — each patient with iron def anemia received an IV syringe of iron sucrose 100 mg every dialysis session for 10 doses

SUMMARY:
the aim of this study is to assess whether increased ferritin after intravenous iron therapy will lead to increased prevalence of major depression among treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. age was above 19 years,
2. patient on maintenance hemodialysis,
3. patient had iron deficiency anemia (ferritin > 100 ng/ml)

Exclusion Criteria:

1. patient has history of depression or already using antidepressant medication,
2. Lack of ferritin level increase ≥ 50% from baseline level before IV iron administration,
3. patient already on oral or intravenous iron supplement

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients with iron deficiency anemia.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Change in patient health questionnaire-9 score | on day 0 of start of intravenous iron and 1 week after completion of intravenous iron
  change in patient health questionnaire-9 score before and after intravenous iron therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hamada, MD, Principal Investigator — Benha University

IPD SHARING:
Plan to Share IPD: No